CLINICAL TRIAL: NCT01945307
Title: Sourcing Human Blood Products to Support the Development of New Vaccines Against Infectious Diseases
Brief Title: Complement 2: Blood Donations to Develop Vaccines Against Infectious Diseases
Acronym: C2
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 2012/11
Record Dates: First submitted 2013-09-13; First posted 2013-09-18 (Estimated); Last update posted 2023-04-04 (Actual); Status verified 2020-10

CONDITIONS: Complement Mediated Bacterial Killing in Healthy Adults
Keywords: Complement; Serum Bactericidal Assay

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum only, no DNA or other blood components are stored.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy adults: Healthy adults aged 18 to 70 years

SUMMARY:
We need human blood to understand the immune response to infection and to test promising new vaccines against infectious diseases in the laboratory. One test is called the Serum Bactericidal Assay (or SBA), which is measure of how effective antibodies are at killing certain bacteria and can be an important measure of how effective a new vaccine may be.

The samples would be used in the laboratory analysis of clinical trials of vaccines used in adults and children, and some samples in pre-clinical (animal) experiments testing new vaccines before they enter human-stage testing. Most people have some form of protection against most bacteria already, so not everyone is a suitable blood donor for this laboratory test. We therefore start by taking a small blood sample and test this one before asking for more blood if we found yours suitable for the work we do.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent for participation in the study
* Aged between 18 and 70 years
* In good health as determined by medical history and clinical judgment of the Investigators
* Able to attend the scheduled visits and to comply with all study procedures
* If found to be a suitable complement that they are willing to be approached for further donations

Exclusion Criteria:

* Body weight less than 50kgs
* Have any known or suspected impairment or alteration of immune function, resulting from, as examples:congenital or acquired immunodeficiency, receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 12 months or long-term systemic corticosteroid therapy, receipt of immunoglobulin or any blood product transfusion within the last 3 months
* Female participants who are pregnant
* Any chronic illness that could, in the opinion of the Investigators, interfere with immune function or with the donation of large volumes of blood (e.g. thrombocytopaenia or coagulopathy, malabsorption disorders, chronic anaemia)
* An individual who is on the delegation log for the study
* Planned blood donation within 4 months of undergoing testing to assess whether the individual is a suitable Complement donor

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adult volunteers, who are willing and able to give informed consent for participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2013-10; Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
To identify healthy adult volunteers whose blood can be used in complement dependent assays | At first visit
  The intrinsic Serum Bactericidal Assay (SBA) of defined infectious bacterial organisms as either a;
  1. complement source with no "intrinsic killing" of defined infectious bacterial organisms
  2. complement source with no killing of defined infectious bacterial organisms following IgG depletion
  3. complement source with "intrinsic killing" of defined infectious bacterial organisms, to act as a positive control

SECONDARY OUTCOMES:
Further exploratory immunology for the development of immunological assays against infectious diseases | At first visit
  To analyse the following in healthy adults;
  * Immunoglobulin G (IgG) antibody concentration against defined target meningococcal, typhoid and shigella strain antigens
  * Complement factor H concentration
  * The relationship between the concentrations of specific anti-meningococcal, anti-typhoid and anti-shigella antibodies and factor H to the ability to mediate intrinsic killing in the SBA assay
  * Any further exploratory immunology to develop laboratory assays measuring the immune responses to vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Pollard, PhD, Principal Investigator — University of Oxford
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine (CCVTM), Oxford, Oxfordshire, United Kingdom

REFERENCES:
- See also: Related Info — http://www.ovg.ox.ac.uk/recruiting-studies